CLINICAL TRIAL: NCT03543917
Title: Post-Stroke Improvement of Motor Function
Acronym: PSIOM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundatia Bio-Forum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSIOM
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-07

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Perfusion

STUDY DESIGN:
Intervention Model Description: The new combination treatment is given to all consecutive patients and compared to literature and between groups (based on the time lapsed between CVA and treatment)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New Medication Combination (Experimental): Intervention: Combination Product: Perfusion with New Combination Medication Intravenous administration of Actovegin, vitamins B1, B6, B12, C, oxytocin/dexamethasone, calcium gluconate, etc in 250 ml normal saline administered during approximately 2 hours
  Interventions: Combination Product: Perfusion with New Combination Medication

INTERVENTIONS:
Combination Product: Perfusion with New Combination Medication — Intravenous administration of Actovegin, vitamins B1, B6, B12, C, oxytocin/dexamethasone, calcium gluconate, etc in 250 ml normal saline administered during approximately 2 hours

SUMMARY:
Open-label clinical study where all new patients presenting with cerebrovascular accidents and consenting to treatment are given intravenously a new combination of medications. Patients are evaluated neurologically with NIHSS scores before treatment administration and at 1 month after the first treatment. Further evaluations at 6 months after treatment by NIHSS and Barthel scores are ongoing

DETAILED DESCRIPTION:
Patients with cerebrovascular accidents (CVA), ischemic (including those with hemorrhagic transformation), are given a new combination of medications which aims to improve neuronal survival, stimulate mitochondrial genesis and the formation of new synapses. This combination is given as an intravenous perfusion with a 2-hr duration and consists of vitamins B1, B6, B12, C, Actovegin, etc.

Before treatment a NIHSS score is given. Each patient receives 3-4 such perfusions in 1 month and afterwards another NIHSS score is obtained.

Patients are monitored afterwards and those who show improvements receive more such treatments, and new NIHSS and Barthel scores are obtained.

Patients are grouped on the basis of the time interval between CVA occurence and first treatment:

* Group 1: 0-35 days
* Group 2: 36-100 days
* Group 3: 101-360 days Improvement of motor function is compared using NIHSS scores between groups, and between literature and groups

ELIGIBILITY:
Inclusion Criteria:

* adults with CVA
* agreeing to treatment in person or by proxy signing of Informed Consent Form
* available for NIHSS evaluation

Exclusion Criteria:

* allergy to any of the substances administered
* scheduled for surgery or other procedures
* not available for NIHSS evaluation after at least 48 hours from treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
NIHSS differential | 1 month after first administration of the combination
  score differential on the National Institutes of Health Stroke Scale(NIHSS); total score is evaluated before treatment and 1 month after first treatment; NIHSS scores range between 0 (best score) and 42 (worst score); the differential quantifies an improvement in neurological function

CONTACTS AND LOCATIONS:
Overall Officials: Felician Stancioiu, Principal Investigator — Fundatia Bio-Forum
Locations (1):
- Fundatia Bio-Forum, Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: No